CLINICAL TRIAL: NCT05273229
Title: Effectiveness of Virtual Gait System Intervention in Motor Function in Older People.
Brief Title: Virtual Gait System Intervention in Older People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1675215UV
Record Dates: First submitted 2022-02-01; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Elderly People
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trail
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Virtual Gait and Physical Exercise (Experimental): Virtual Gait and Physical Exercise Virtual Gait The subject will be stand up with a standing opposite a mirror (from the waist up) and a screen (from the waist down) where a video of treadmill gait of a person will be projected.
  Physical Exercise Specific gait exercise was conducted.
  Interventions: Other: Virtual Gait; Other: Physical exercise
- Documental projection and Physical Exercise (Sham Comparator): Physical Exercise Specific gait exercise was conducted.
  Documental projection The subject will be stand up with a standing opposite a mirror (from the waist up) and a screen (from the waist down) where video without any type of animal or human movement was showed.
  Interventions: Other: Physical exercise; Other: Sham Virtual Gait
- Virtual Gait (Experimental): only the virtual gait program will be carried out, detailed in Arm I.
  Interventions: Other: Virtual Gait
- Virtual Gait Sham (Sham Comparator): Documental projection The subject will be stand up with a standing opposite a mirror (from the waist up) and a screen (from the waist down) where video without any type of animal or human movement was showed.
  Interventions: Other: Sham Virtual Gait

INTERVENTIONS:
Other: Virtual Gait — Virtual Gait: the patient will be placed in a standing position (with an ad-hoc designed help system) in front of a mirror (from the waist up) and a screen (from the waist down) where a video of legs walking on a treadmill will be projected and overcoming obstacles. Projected legs will be customized based on height, using the tibia length method.
  Arms: Virtual Gait; Virtual Gait and Physical Exercise
Other: Physical exercise — PE: it will be divided into two parts: in the first one, a gait technique training will be carried out and, in the second, a leg strength training, for 30 min. Exercises:
  * Coordination exercises: normal and lateral parallel walking and walking with obstacles.
  * Functional exercises such as climbing stairs, etc.
  * Lower limb strength exercises. Strength exercises will be prescribed according to the guidelines of the American College of Sports Medicine (ACSM). Progression will be customized based on individual abilities.
  Arms: Documental projection and Physical Exercise; Virtual Gait and Physical Exercise
Other: Sham Virtual Gait — only the placebo virtual gait.
  Arms: Documental projection and Physical Exercise; Virtual Gait Sham

SUMMARY:
Previous studies have shown that the neuroplasticity of the residual corticospinal fibers, the motor cortex and the spinal neurons plays an important role in the spontaneous functional recovery of people with neurological or musculoskeletal pathology. However, it is also possible to stimulate the neuroplasticity mechanisms of these structures through techniques aimed at rehabilitating different deficits (for example, motor function or sensitivity). In general, intervention programs are usually carried out, in most cases, using low-cost strategies such as therapeutic physical exercise programs.

The objective of this study is to analyze the effectiveness of visual illusion therapies in combination with conventional exercises on the symptoms and signs related to elderly people.

The study will include the realization of three measurements that will be carried out one day before starting the program, one day after finishing it, and one month later (follow-up).

The clinical assessment will be composed of the study of the following variables: Motor function and motor skills, Upper limb isometric force, Muscle activation, Muscle tone, Quality of life, Functionality. All interventions will last eight weeks and will be planned according to the availability of volunteers. In each session, it will be recorded if any type of adverse effect occurs. There will be four types of interventions: i. Visual Illusion (IV) and therapeutic exercise program (PE), ii.placebo and PE, iii. IV, iv. IV placebo.

DETAILED DESCRIPTION:
The prevalence of gait and balance disorders increases by 10% between 60 and 69 years of age, reaching 60% in people over 80 years of age or 82% in people over 85 years of age. These disorders are also characteristic of populations with different neurological or musculoskeletal conditions. This supposes a profound psychological and socioeconomic impact on the affected person's life, in addition to the implicit physical impact.

After an injury (whether acquired or due to deterioration due to aging), there is a spontaneous functional recovery that can have different paths depending on the characteristics of the injury and the person. Previous studies have shown that the neuroplasticity of residual corticospinal fibers, motor cortex and spinal neurons plays an important role in the spontaneous functional recovery of people with neurological or musculoskeletal pathology, as well as in the reorganization of the spinal system. motor skills of the elderly. However, it is also possible to stimulate the neuroplasticity mechanisms of these structures through techniques aimed at rehabilitating different deficits (for example, motor function or sensitivity). In general, intervention programs aimed at improving neuroplasticity are usually carried out, in most cases, using low-cost strategies such as therapeutic physical exercise programs.

This nerve reorganization and recovery can also be influenced by the activity of mirror neurons, which are found in motor and premotor areas and also in other cortical and subcortical areas; and report activation when they observe an action with a specific purpose. The activity of these neurons has been studied in different populations with Central Nervous System (CNS) involvement, such as strokes, head injuries, Parkinson's or Alzheimer's. For its study, experimental investigations have been carried out applying different interventions that modify the activity of mirror neurons, such as mirror therapy, virtual reality therapies, Action-Observation therapies or visual illusion. In general, promising results have been obtained in all these populations, except in the case of advanced-stage Alzheimer's disease.

Visual illusion therapies have been used in different populations, such as spinal cord injury, with promising results. However, this type of therapy has not been studied in other populations with different neurological or musculoskeletal conditions, as well as in the elderly population.

The main objective of this study is to evaluate the efficacy of a virtual walking treatment (visual illusion) comparing it with interventions combined with specific physical exercise of walking in elderly people, on the functional capacity of this population.

Taking all of the above into account, the main objective of this study is to evaluate the efficacy of a virtual gait treatment (visual illusion) compared to interventions combined with specific physical gait exercise in people with disabilities or older people, on functional capacity of these populations. Specifically, it is intended to know the impact of virtual gait therapy on:

* The actual gait, both speed and resistance.
* Functionality in mobility activities and postural control.
* Isometric strength of lower extremities.
* Muscular tone, stiffness and elasticity of the leg muscles.
* Neuropathic pain and sensitivity.

Therefore, this study aims to provide knowledge to the scientific community on how the mechanisms of neuroplasticity and specifically mirror neurons can influence the rehabilitation of people with disabilities and the elderly and, in addition, to propose a specific treatment methodology for the rehabilitation of the march in this type of population.

The recruitment and execution of the interventions will be carried out in a room set up within the Faculty of Physiotherapy of the University of Valencia. All procedures will be carried out under the principles of the Declaration of Helsinki (World Medical Association) and will be approved by the ethics committee of the University of Valencia. In addition, all participants will be asked to sign an informed consent that will include all the sections required by this committee.

A minimum of 20 participants per group is established, establishing a power of 80%, an ability to detect a small effect size (Cohen's d = 0.3) for the main variable resistance measured with the 2min Walking Test and a probability of type error. I of 0.05, resulting in a total of 80 participants. In order to minimize possible losses, 25% more patients per group will be added, so 100 people will participate in the study.

The study will contemplate the realization of three measurements that will be carried out one day before starting the program, one day after finishing it, and 1 month later. These will be carried out by team members who are blind to the assignment of the interventions.

In the first evaluation, anthropometric and demographic data will be collected (i.e. height, weight, age, educational level, possible comorbidities, etc.) with the aim of controlling, if necessary, these confounding variables.

The data analysis will be carried out using the SPSS statistical program (version 26). The normality of the sample will be analyzed using the Shapiro Wilk test and homoscedasticity using the Levene test. For the comparison between groups, a mixed factorial ANOVA will be used, and for the comparison between pairs of groups the Bonferroni correction will be used. In the event that there may be a confounding factor that meets the requirements to be analyzed as a covariate, an ANCOVA will be used. Statistically significant differences will be assumed when the p-value is less than 0.05.

All interventions will last eight weeks and will be planned according to the availability of volunteers. In each session, it will be recorded if any type of adverse effect occurs.

There will be four types of interventions resulting of a combination of:

Visual Illusion (IV): the patient will be placed in a standing position (with a help system designed ad-hoc) in front of a mirror (from the waist up) and a screen (from the waist down) where a video of legs walking will be projected. a treadmill and overcoming obstacles.. This program will last 10 minutes.

Therapeutic exercise program (PE): Physical exercise program for the lower extremities will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Mini-Mental State Examination >23 points.
* Ability to walk with or without aids

Exclusion Criteria:

* Lower limbs traumatic pathology.
* Other nervous system alterations.
* Vestibular diseases.
* Other diseases.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Walking distance (meters) | 2 minutes
  2 min walk test
Functionality | 10 minutes
  FallSkip
Muscular tone | 10 minutes
  MyotonPRO
Lower extremity functionality | 10 minutes
  Physical performance with Short Physical Performance Battery (SPPB). It is an assessment tool for evaluation of lower extremity functioning in older persons.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy Recruiting Valencia, Spain, 46010, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Mahlknecht P, Kiechl S, Bloem BR, Willeit J, Scherfler C, Gasperi A, Rungger G, Poewe W, Seppi K. Prevalence and burden of gait disorders in elderly men and women aged 60-97 years: a population-based study. PLoS One. 2013 Jul 24;8(7):e69627. doi: 10.1371/journal.pone.0069627. Print 2013. PMID 23894511
- [Background] Sudarsky L. Gait disorders: prevalence, morbidity, and etiology. Adv Neurol. 2001;87:111-7. No abstract available. PMID 11347214
- [Background] Nguyen L, Murphy K, Andrews G. Cognitive and neural plasticity in old age: A systematic review of evidence from executive functions cognitive training. Ageing Res Rev. 2019 Aug;53:100912. doi: 10.1016/j.arr.2019.100912. Epub 2019 May 30. PMID 31154013
- [Background] Aitkens M. A legacy of surgeons. Minn Med. 1988 Oct;71(10):592-6. No abstract available. PMID 3070327
- [Background] Jeannerod M. The hand and the object: the role of posterior parietal cortex in forming motor representations. Can J Physiol Pharmacol. 1994 May;72(5):535-41. doi: 10.1139/y94-077. PMID 7954083
- [Background] Dushanova J, Donoghue J. Neurons in primary motor cortex engaged during action observation. Eur J Neurosci. 2010 Jan;31(2):386-98. doi: 10.1111/j.1460-9568.2009.07067.x. Epub 2010 Jan 13. PMID 20074212
- [Background] Vigneswaran G, Philipp R, Lemon RN, Kraskov A. M1 corticospinal mirror neurons and their role in movement suppression during action observation. Curr Biol. 2013 Feb 4;23(3):236-43. doi: 10.1016/j.cub.2012.12.006. Epub 2013 Jan 3. PMID 23290556
- [Background] Onishi H. [The current status and future of prosthetic joint replacement]. Kango Gijutsu. 1988 Oct;34(13):1566-71. No abstract available. Japanese. PMID 3210396